CLINICAL TRIAL: NCT01149772
Title: Cognitive Behavioral Therapy in Primary Care: Treating the Medically Ill
Brief Title: Adjusting to Chronic Conditions Using Education, Support, and Skills
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 09-088; 2619 (Other Grant/Funding Number: HSR-D)
Record Dates: First submitted 2010-06-10; First posted 2010-06-23 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Heart Failure; Anxiety; Depression
Keywords: Chronic Obstructive Pulmonary Disease; Heart Failure; Anxiety; Depression
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACCESS (Experimental): Medically ill patients received six-sessions of cognitive behavioral therapy tailored to their unique needs. Patients received 2 core modules and 3 elective modules. Elective modules focused on physical health, cognitive restructuring, behavioral activation, and relaxation. The six session was a wrap up that everyone received. Patients also had the option to receive 2 follow-up booster sessions to aid in maintenance of skills learned.
  Interventions: Behavioral: ACCESS
- Enhanced Usual Care (No Intervention): Patients in this arm received feedback about their physical and emotional health functioning and were still able to receive usual primary care services.

INTERVENTIONS:
Behavioral: ACCESS — Participants received 6 treatment sessions (2 core and 4 electives). The two core modules are increasing awareness and controlling physical and emotional symptoms. After completion of the core modules the participant was able to choose elective modules from Managing Physical Health, The Power of Thoughts, Increasing Pleasant Activities, and Relaxation. Participants were required to complete the first session in person and subsequent sessions participants had the option to complete in-person or over the phone. Participants also had the option to receive 2 brief follow-up booster calls to aid in reinforcing the changes made.
  Arms: ACCESS

SUMMARY:
The current study seeks to test the effectiveness of a talk-therapy intervention designed to better meet the needs of chronically ill Veterans. This project looks to recruit 450 Veterans with either chronic obstructive pulmonary disease (COPD) or heart failure (HF) who also have symptoms of worry, stress, anxiety, or sadness. Participants will be randomly put into either the talk-therapy intervention or enhanced usual care.

The talk therapy intervention will be provided by VA clinicians in the primary care setting and will consist of 6 core meetings (30-45 minutes in duration) and 2 follow-up telephone meetings. Enhanced usual care participants will receive feedback regarding the assessment findings and educational materials on COPD and/or HF, depression and anxiety.

DETAILED DESCRIPTION:
Diseases of the heart and circulatory system, namely, Chronic Obstructive Pulmonary Disease (COPD) and Heart Failure (HF), are two of the most common and disabling chronic diseases. Both COPD and HF account for significant disability, mortality, and healthcare costs and are associated with lower health status and more functional and social limitations than other chronic illnesses, such as hypertension and diabetes. As our population ages and life span increases, the numbers of patients with these conditions and the subsequent healthcare costs will increase dramatically.

The symptoms associated with COPD and HF can significantly affect daily functioning. Physical symptoms are often linked to increased levels of psychological distress, namely, anxiety and depression, which significantly affect quality of life and functioning above and beyond the impact of the medical disease. As depression and anxiety are modifiable clinical factors, there is a potential to significantly alter patient outcomes, as well as use of healthcare services. However, focused interventions are needed, given the high risk for poor mental health treatment and underuse of mental health services in persons with COPD and HF. Unfortunately, few intervention studies have been conducted in medically ill patients with these conditions. The current project will examine whether existing VA clinicians in the primary care setting, with training and support, can effectively administer a structured Cognitive Behavioral Therapy (CBT) intervention for depressed and anxious Veterans with COPD and HF.

ELIGIBILITY:
Inclusion Criteria:

* COPD and/or HF diagnosis; confirmation based upon medical chart review.
* clinically significant symptoms for anxiety and/or depression.

Exclusion Criteria:

* cognitive impairment
* presence of bipolar, psychotic or substance abuse disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2011-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Cully, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (2):
- United States (2):
  - VA Medical Center, Oklahoma City, Oklahoma City, Oklahoma
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

REFERENCES:
- [Result] Mignogna J, Hundt NE, Kauth MR, Kunik ME, Sorocco KH, Naik AD, Stanley MA, York KM, Cully JA. Implementing brief cognitive behavioral therapy in primary care: A pilot study. Transl Behav Med. 2014 Jun;4(2):175-83. doi: 10.1007/s13142-013-0248-6. PMID 24904701
- [Result] Cully JA, Curry AD, Ryan SR, Malik A, Zeno D, Willcockson IU. Development of a computer-aided training program for brief cognitive-behavioral therapy in primary care. Acad Psychiatry. 2013 Mar 1;37(2):120-4. doi: 10.1176/appi.ap.11040078. No abstract available. PMID 23475245
- [Result] Cully JA, Armento ME, Mott J, Nadorff MR, Naik AD, Stanley MA, Sorocco KH, Kunik ME, Petersen NJ, Kauth MR. Brief cognitive behavioral therapy in primary care: a hybrid type 2 patient-randomized effectiveness-implementation design. Implement Sci. 2012 Jul 11;7:64. doi: 10.1186/1748-5908-7-64. PMID 22784436
- [Result] Mignogna J, Cully J. Depression and Anxiety in Patients with COPD: A Focus on Psychological Treatments in Ambulatory Care Settings. Current respiratory medicine reviews. 2012 Apr 1; 8(2):137-144(8).
- [Result] Hundt NE, Bensadon BA, Stanley MA, Petersen NJ, Kunik ME, Kauth MR, Cully JA. Coping mediates the relationship between disease severity and illness intrusiveness among chronically ill patients. J Health Psychol. 2015 Sep;20(9):1186-95. doi: 10.1177/1359105313509845. Epub 2013 Dec 1. PMID 24296739
- [Result] Breland JY, Hundt NE, Barrera TL, Mignogna J, Petersen NJ, Stanley MA, Cully JA. Identification of Anxiety Symptom Clusters in Patients with COPD: Implications for Assessment and Treatment. Int J Behav Med. 2015 Oct;22(5):590-6. doi: 10.1007/s12529-014-9450-2. PMID 25622813
- [Derived] Hundt NE, Renn BN, Sansgiry S, Petersen NJ, Stanley MA, Kauth MR, Naik AD, Kunik ME, Cully JA. Predictors of response to brief CBT in patients with cardiopulmonary conditions. Health Psychol. 2018 Sep;37(9):866-873. doi: 10.1037/hea0000595. PMID 30138022
- [Derived] Mignogna J, Martin LA, Harik J, Hundt NE, Kauth M, Naik AD, Sorocco K, Benzer J, Cully J. "I had to somehow still be flexible": exploring adaptations during implementation of brief cognitive behavioral therapy in primary care. Implement Sci. 2018 Jun 5;13(1):76. doi: 10.1186/s13012-018-0768-z. PMID 29866141
- [Derived] Renn BN, Hundt NE, Sansgiry S, Petersen NJ, Kauth MR, Kunik ME, Cully JA. Integrated Brief Cognitive Behavioral Therapy Improves Illness Intrusiveness in Veterans With Chronic Obstructive Pulmonary Disease. Ann Behav Med. 2018 Jul 13;52(8):686-696. doi: 10.1093/abm/kax045. PMID 29860524
- [Derived] Thakur ER, Sansgiry S, Petersen NJ, Stanley M, Kunik ME, Naik AD, Cully JA. Cognitive and Perceptual Factors, Not Disease Severity, Are Linked with Anxiety in COPD: Results from a Cross-Sectional Study. Int J Behav Med. 2018 Feb;25(1):74-84. doi: 10.1007/s12529-017-9663-2. PMID 28779469
- [Derived] Cully JA, Stanley MA, Petersen NJ, Hundt NE, Kauth MR, Naik AD, Sorocco K, Sansgiry S, Zeno D, Kunik ME. Delivery of Brief Cognitive Behavioral Therapy for Medically Ill Patients in Primary Care: A Pragmatic Randomized Clinical Trial. J Gen Intern Med. 2017 Sep;32(9):1014-1024. doi: 10.1007/s11606-017-4101-3. Epub 2017 Jun 20. PMID 28634906

RESULTS

PARTICIPANT FLOW:
Groups:
- ACCESS: Adjusting to Chronic Conditions Using Education, Support, and Skills: Participants in this condition will receive 6 active weekly treatment sessions (2 core and 4 electives). The two core modules are increasing awareness and controlling physical and emotional symptoms. After completion of the core modules the participant will be able to choose elective modules from Managing your Physical Health, The Power of Thoughts, Increasing Pleasant Activities, and Learning How to Relax. Participants are required to complete the first session in person Subsequent sessions participants have the option to complete in-person or over the phone. After completion of the active treatment sessions, the participant can receive 2 brief follow-up booster calls to aid in reinforcing the skills learned.
- Enhanced Usual Care: Patients in this arm receive feedback about their physical and emotional health functioning and subsequently receive usual primary care services.
Period: Overall Study
Arm/Group | ACCESS | Enhanced Usual Care
Started | 180 | 122
Completed | 132 | 101
Not Completed | 48 | 21

BASELINE CHARACTERISTICS:
Population: This is the total number of participants eligible after baseline and were randomized into each arm.
Groups:
- ACCESS: Adjusting to Chronic Conditions Using Education, Support, and Skills: Participants in this condition will receive 6 active weekly treatment sessions (2 core and 4 electives). The two core modules are increasing awareness and controlling physical and emotional symptoms. After completion of the core modules the participant will be able to choose elective modules from Managing your Physical Health, The Power of Thoughts, Increasing Pleasant Activities, and Learning How to Relax. After completion of the active treatment sessions, the participant will receive 2 brief follow-up booster calls. The follow up calls provide the opportunity for the participant to review skills learned, address any questions or difficulties, and reinforce changes made. Each active treatment session lasts 30 - 40 minutes and the booster calls last 10 - 15 minute.
- Total: Total of all reporting groups
Arm/Group | ACCESS | Enhanced Usual Care | Total
Number analyzed (Participants) | 180 | 122 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (8.8) | 66.5 (8.3) | 65.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 168 | 116 | 284
Region of Enrollment [Number; unit: participants]
  United States | 180 | 122 | 302
Patient Health Questionnaire (PHQ9) [Mean (Standard Deviation); unit: units on a scale] — The PHQ9 measures an individual's level of depression. The measure is summed and ranges from 0 - 27 (individual item score range 0 - 3 per 9 items); where higher scores = worse symptoms.
  units on a scale | 13.8 (4.6) | 14.9 (5.0) | 14.2 (4.8)
Beck Anxiety Inventory (BAI) [Mean (Standard Deviation); unit: units on a scale] — The BAI measures an individual's level of anxiety. The measure is summed and ranges from 0 - 63 (individual item score range 0 - 3 per 21 items); where higher scores = worse symptoms.
  units on a scale | 21.4 (8.9) | 22.9 (10.7) | 22.0 (9.6)
Chronic Respiratory Questionnaire_Mastery [Mean (Standard Deviation); unit: units on a scale] — The CRQ measures the quality of life of patients with a chronic respiratory disease. The subscale Mastery looks at the patients perceived control over the condition. The CRQ is a mean score and ranges from 1 - 7, where a higher score = better health.
  units on a scale | 3.63 (1.03) | 3.48 (1.16) | 3.57 (1.08)
Chronic Respiratory Questionnaire_Dyspnea [Mean (Standard Deviation); unit: units on a scale] — The CRQ measures the quality of life of patients with a chronic respiratory disease. The subscale Dyspnea looks at how much shortness of breath a patient experiences. The CRQ is a mean score and ranges from 1 - 7, where a higher score = better health.
  units on a scale | 3.05 (.95) | 2.90 (1.03) | 2.99 (.98)
Chronic Respiratory Questionnaire_Fatigue [Mean (Standard Deviation); unit: units on a scale] — The CRQ measures the quality of life of patients with a chronic respiratory disease. This subscale measures the amount of fatigue patients experience with the condition. The CRQ is a mean score and ranges from 1 - 7, where a higher score = better health.
  units on a scale | 2.63 (.90) | 2.43 (.97) | 2.55 (.93)
Kansas City Cardiomyopathy Questionnaire (KCCQ) [Mean (Standard Deviation); unit: units on a scale] — The KCCQ measures the health status of patients with congestive heart failure. The overall score is a mean score scaled from 0 - 100; where 0 represents most severe/limited functioning.
  units on a scale | 36.93 (14.94) | 37.03 (19.36) | 36.97 (16.81)

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire -9 (PHQ-9)
Description: The PHQ-9 measures an individual's level of depression. The measure is summed and ranges from 0 - 27 (individual item score range 0 - 3 per 9 items); where higher scores = worse symptoms.
Time Frame: 4 month (post treatment), 8 month follow/up, and 12 month follow/up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACCESS | Enhanced Usual Care
Number analyzed (Participants) | 132 | 101
units on a scale
  4 Month | 10.35 (5.08) | 13.28 (5.82)
  8 Month | 10.32 (5.48) | 13.49 (6.05)
  12 Month | 10.59 (5.07) | 13.22 (6.38)

2. Primary Outcome: Beck Anxiety Inventory (BAI)
Description: The BAI measures an individual's level of anxiety. The measure is summed and ranges from 0 - 63 (individual item score range 0 -3 per 21 items); were higher scores = worse symptoms.
Time Frame: 4 month (post treatment), 8 month follow/up, and 12 month follow/up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACCESS | Enhanced Usual Care
Number analyzed (Participants) | 132 | 101
units on a scale
  4 Month | 17.42 (8.52) | 22.67 (11.18)
  8 Month | 16.85 (9.27) | 21.59 (11.41)
  12 Month | 16.97 (7.91) | 21.19 (11.40)

3. Primary Outcome: Chronic Respiratory Questionnaire_Fatigue
Description: The Chronic Respiratory Questionnaire (CRQ) measures the quality of life of patients with a chronic respiratory disease. This subscale measures the amount of fatigue patients experience with the condition. The CRQ is a mean score and ranges from 1 - 7, where a higher score = better health.
Time Frame: 4 month (post treatment), 8 month follow/up, 12 month follow/up
Population: Only patients experiencing chronic lung problems (COPD, emphysema, bronchitis, asthma) completed this assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ACCESS: Adjusting to Chronic Conditions Using Education, Support, and Skills: Participants in this condition will receive 6 active weekly treatment sessions (2 core and 4 electives). The two core modules are increasing awareness and controlling physical and emotional symptoms. After completion of the core modules the participant will be able to choose elective modules from Managing your Physical Health, The Power of Thoughts, Increasing Pleasant Activities, and Learning How to Relax. Participants are required to complete the first session in person Subsequent sessions participants have the option to complete in-person or over the phone. After completion of the active treatment sessions, the participant can receive 2 brief follow-up booster calls. The follow up calls provide the opportunity for the participant to review skills learned, address any questions or difficulties, and reinforce changes made.
Arm/Group | ACCESS | Enhanced Usual Care
Number analyzed (Participants) | 101 | 74
units on a scale
  4 month | 3.20 (1.08) | 2.58 (1.08)
  8 month | 3.11 (1.09) | 2.68 (1.01)
  12 month | 3.05 (1.06) | 2.77 (1.15)

4. Primary Outcome: Chronic Respiratory Questionnaire_Mastery
Description: The Chronic Respiratory Questionnaire (CRQ) measures the quality of life of patients with a chronic respiratory disease. The subscale Mastery looks at the patient's perceived control over the condition. The CRQ is a mean score and ranges from 1 - 7, where a higher score = better health
Time Frame: 4 month (post treatment), 8 month follow/up, 12 month follow/up
Population: Only patients experiencing chronic lung problems (COPD, emphysema, bronchitis, asthma) completed this assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACCESS | Enhanced Usual Care
Number analyzed (Participants) | 101 | 74
units on a scale
  4 month | 4.25 (1.14) | 3.51 (1.19)
  8 month | 4.20 (1.20) | 3.45 (1.22)
  12 month | 3.96 (1.11) | 3.62 (1.28)

5. Primary Outcome: Chronic Respiratory Questionnaire_Dyspnea
Description: The Chronic Respiratory Questionnaire (CRQ) measures the quality of life of patients with a chronic respiratory disease. The subscale Dyspnea looks at how much shortness of breath a patient experiences. The CRQ is a mean score and ranges from 1 - 7, where a higher score = better health.
Time Frame: 4 month (post treatment), 8 month follow/up, 12 month follow/up
Population: Only patients experiencing chronic lung problems (Chronic Obstructive Pulmonary Disease, emphysema, bronchitis, asthma) completed this assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACCESS | Enhanced Usual Care
Number analyzed (Participants) | 101 | 74
units on a scale
  4 month | 3.37 (1.15) | 2.94 (.98)
  8 month | 3.27 (1.02) | 3.03 (.89)
  12 month | 3.07 (.99) | 3.11 (1.05)

6. Primary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: The KCCQ measures the health status of patients with congestive heart failure. The overall score is a mean score scaled from 0 - 100; where 0 represents most severe/limited functioning.
Time Frame: 4 month (post treatment), 8 month follow/up, and 12 month follow/up
Population: Only patients randomized for heart failure was required to complete the assessment. There were fewer patients randomized for congestive heart failure (CHF) as compared to COPD.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACCESS | Enhanced Usual Care
Number analyzed (Participants) | 46 | 40
units on a scale
  4 month | 40.25 (15.12) | 41.81 (19.21)
  8 month | 41.34 (19.89) | 36.23 (18.21)
  12 month | 42.89 (18.30) | 41.68 (20.81)

ADVERSE EVENTS:
Time Frame: Data on Adverse events was collected for a period of 1 year. This is the length of time participants were in the study.
Description: Although there were adverse events during the course of the study, none were determined to be related to the study.
Groups:
- ACCESS: ACCESS: Participants received 6 treatment sessions (2 core and 4 electives). The two core modules are increasing awareness and controlling physical and emotional symptoms. After completing core modules the participant was able to choose elective modules from Managing Physical Health, The Power of Thoughts, Increasing Pleasant Activities, and Relaxation. Participants were required to complete the first session in person and subsequent sessions participants had the option to complete in-person or over the phone. After completion of the active treatment sessions, the participant can receive 2 brief follow-up booster calls to aid in reinforcing the skills learned.
Arm/Group | ACCESS | Enhanced Usual Care
Serious Adverse Events (participants affected / at risk) | 8/180 | 9/122
Other Adverse Events (participants affected / at risk) | 57/180 | 52/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACCESS (N=180) | Enhanced Usual Care (N=122)
Death (Investigations) | 4 | 5 — These deaths were determined not to be related to the study.
Hospitalizations (Cardiac disorders) | 4 | 4 — These adverse events were determined not to be related to the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACCESS (N=180) | Enhanced Usual Care (N=122)
Depression (Psychiatric disorders) | 33 | 24 — Patient eligibility was based on elevated symptoms of depression. Patients were monitored for significant increases in depression symptoms. No known adverse events were attributable to the study.
Anxiety (Psychiatric disorders) | 24 | 28 — Patient eligibility was based on elevated symptoms of anxiety. Patients were monitored for significant increases in anxiety symptoms. No adverse events were known to be attributable to the study.

LIMITATIONS AND CAVEATS:
There were some deaths and hospitalizations during the study, however, none of the adverse events reported were determined to be related to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes